CLINICAL TRIAL: NCT01105273
Title: HLA-haploidentical Allogeneic Hematopoietic Cell Transplantation Using CD3±CD19 Depletion for Patients With Aplastic Anemia After Conditioning of Fludarabine, Cyclophosphamide and Antithymocyte Globulin
Brief Title: Human Leukocyte Antigen (HLA)-Haploidentical Hematopoietic Stem Cell Transplantation for Patients With Aplastic Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Joon Im, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCPHO-SCT0802
Record Dates: First submitted 2010-04-08; First posted 2010-04-16 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Aplastic Anemia
Keywords: Aplastic anemia; Fludarabine; CD3±CD19 depletion; Haploidentical hematopoietic stem cell transplantation
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum; Filgrastim; fludarabine; Cyclophosphamide

ARMS (1):
- HAPLO (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: CD3±CD19 depleted hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin — On days -3 to -1
Biological: filgrastim — Beginning on day 4 and continuing until blood counts recover
Drug: Fludarabine — 30mg/M2 once daily IV on days -6 to -2
Drug: Cyclophosphamide — 60 mg/kg IV on day-3 and -2
Procedure: CD3±CD19 depleted hematopoietic stem cell transplantation — Immunogenetic depletion on CliniMACS

SUMMARY:
Rationale: Chemotherapy with fludarabine, cyclophosphamide and anti-thymocyte globulin may induce the engraftment cross the immunologic barrier in the setting of HLA-haploidentical allogeneic hematopoietic cell transplantation. In addition, depletion CD3±CD19 cells may contribute to prevent developing severe acute graft versus host disease (GVHD) in haploidentical transplantation.

Purpose: This phase I/II trial is to evaluate the safety and efficacy of fludarabine, cyclophosphamide and antithymocyte globulin with CD3±CD19 depleted graft from haploidentical donors in treating patients with aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of life-threatening marrow failure (severe aplastic anemia) of nonmalignant etiology meeting 2 of the following criteria:

  * Granulocyte count < 500/mm3,
  * Corrected reticulocyte count < 1%,
  * Platelet count < 20,000/mm3
* No HLA-identical family member or closely matched (8 of 8 HLA-locus match) unrelated marrow donor available
* HLA-haploidentical related donor available

Exclusion Criteria:

* Paroxysmal nocturnal hemoglobinuria or Fanconi anemia
* Clonal cytogenetic abnormalities or myelodysplastic syndromes
* Active fungal infections
* HIV positive
* Severe disease other than aplastic anemia that would severely limit the probability of survival during the graft procedure
* Pregnant or nursing

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To assess the engraftment rate and survival of CD3±CD19 depleted haploidentical peripheral blood stem cell transplantation after conditioning with fludarabine, cyclophosphamide and anti-thymocyte globulin. | 2 years post-transplant

SECONDARY OUTCOMES:
To assess engraftment and graft failure | 28 days post-transplant
  Number of patients who failed to engraft by 28 days.
To estimate the risk of acute GVHD | 100 days post-transplant
  Number of patients with acute GVHD.
To assess treatment related mortality | 100 days post-transplant
  Number of death after transplantation
To estimate overall survival | 1 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Ho Joon Im, MD & PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Woodard P, Cunningham JM, Benaim E, Chen X, Hale G, Horwitz E, Houston J, Kasow K, Leung W, Wang W, Yusuf U, Handgretinger R. Effective donor lymphohematopoietic reconstitution after haploidentical CD34+-selected hematopoietic stem cell transplantation in children with refractory severe aplastic anemia. Bone Marrow Transplant. 2004 Feb;33(4):411-8. doi: 10.1038/sj.bmt.1704358. PMID 14676782
- [Background] Kremens B, Basu O, Grosse-Wilde H, Sauerwein W, Schaefer UW, Havers W. Transplantation of CD34-enriched peripheral stem cells from an HLA-haplotype mismatched donor to a patient with severe aplastic anemia. Bone Marrow Transplant. 2001 Jan;27(1):111-3. doi: 10.1038/sj.bmt.1702748. PMID 11244448
- [Background] Lacerda JF, Martins C, Carmo JA, Lourenco F, Juncal C, Ismail S, Lacerda JM. Haploidentical stem cell transplantation with purified CD34+ cells after a chemotherapy-alone conditioning regimen in heavily transfused severe aplastic anemia. Biol Blood Marrow Transplant. 2005 May;11(5):399-400. doi: 10.1016/j.bbmt.2005.02.007. No abstract available. PMID 15846294
- [Background] Klingebiel T, Cornish J, Labopin M, Locatelli F, Darbyshire P, Handgretinger R, Balduzzi A, Owoc-Lempach J, Fagioli F, Or R, Peters C, Aversa F, Polge E, Dini G, Rocha V; Pediatric Diseases and Acute Leukemia Working Parties of the European Group for Blood and Marrow Transplantation (EBMT). Results and factors influencing outcome after fully haploidentical hematopoietic stem cell transplantation in children with very high-risk acute lymphoblastic leukemia: impact of center size: an analysis on behalf of the Acute Leukemia and Pediatric Disease Working Parties of the European Blood and Marrow Transplant group. Blood. 2010 Apr 29;115(17):3437-46. doi: 10.1182/blood-2009-03-207001. Epub 2009 Dec 29. PMID 20040760
- [Result] Koh KN, Im HJ, Kim BE, Choi ES, Jang S, Kwon SW, Park CJ, Seo JJ. Haploidentical haematopoietic stem cell transplantation using CD3 or CD3/CD19 depletion and conditioning with fludarabine, cyclophosphamide and antithymocyte globulin for acquired severe aplastic anaemia. Br J Haematol. 2012 Apr;157(1):139-42. doi: 10.1111/j.1365-2141.2011.08924.x. Epub 2011 Nov 5. No abstract available. PMID 22055111
- [Derived] Im HJ, Koh KN, Suh JK, Lee SW, Choi ES, Jang S, Kwon SW, Park CJ, Seo JJ. Refinement of treatment strategies in ex vivo T-cell-depleted haploidentical SCT for pediatric patients. Bone Marrow Transplant. 2015 Feb;50(2):225-31. doi: 10.1038/bmt.2014.232. Epub 2014 Oct 13. PMID 25310303
- See also: Anemia — http://www.nlm.nih.gov/medlineplus/anemia.html
- See also: Fludarabine — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=021679141&QV1=FLUDARABINE
- See also: Cyclophosphamide — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet